CLINICAL TRIAL: NCT06765122
Title: Program for Alleviating and Reducing Trauma and Stress for Intimate Partner Violence
Acronym: PARTS-IPV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Washington State Department of Social and Health Services (Other); Washington State Department of Commerce Office of Crime Victims Advocacy (Unknown); Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHA-IRB-24-25-352
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Interpersonal Violence
Keywords: Interpersonal Violence, domestic violence; Program For Alleviating Relationship Trauma and Stress; Internal Family Systems (IFS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PARTS-NB (Experimental): All study participants will be in the PARTS-NB arm and go through the treatment program called "Program for Alleviating Relationship Trauma and Stress through New Behaviors".
  Interventions: Behavioral: Program for Alleviating Relationship Trauma and Stress through New Behaviors (PARTS-NB)

INTERVENTIONS:
Behavioral: Program for Alleviating Relationship Trauma and Stress through New Behaviors (PARTS-NB) — PARTS-NB (Program For Alleviating Relationship Trauma and Stress through New Behaviors) is a group-based program for people who use violence and aggression in intimate relationships. Phase I is 4-weeks of 120 minutes of weekly group-based sessions focused on clarifying the way parts work in the mind, increasing inner compassion and emotion regulation, and explaining the role of trauma and stress in substance use and the use of violence in relationships. Phase II lasts 8-weeks, maintaining the 120 minutes of weekly group-based sessions. This phase introduces the model and focuses on practicing "unblending," helping individuals gain awareness and acceptance of internal and external experiences. The final phase, Phase III runs 8 weeks and consists of weekly 120-minute group sessions which addresses and releases trauma-based beliefs and experiences through a process called "unburdening."
  Other Names: PARTS-IPV

SUMMARY:
This research study investigates the feasibility and acceptability of a group-based treatment program for reducing stress, trauma, substance use, and use of violence among individuals who were court-mandated to attend a program after committing an act(s) of domestic violence.

DETAILED DESCRIPTION:
Our program is adapted from the original PARTS (Program For Alleviating and Reducing Trauma and Stress). And will include unique and specific elements for People who Use Violence (PUV) in intimate relationships. PARTS-IPV is structured in three phases. Phase I is 4-weeks of 120 minutes of weekly group-based sessions. This phase introduces the model and creates a "brave container" to address any ambivalence towards the program. Phase II lasts 8-weeks, maintaining the 120 minutes of weekly group-based sessions. This second phase focuses on "unblending" through working with Parts and connecting with Self. The final phase, Phase III runs 8 weeks and consists of weekly 120-minute group sessions focused "unburdening". Throughout the intervention, individual sessions will be help with an IFS-trained clinician at a frequency of around once a month for a total of 6 individual sessions. These sessions will focus on enhancing group participation, providing space for trauma counseling and unburdening, addressing negative beliefs or concerns that may arise about group, and providing insights into person reasons for the use of violence in intimate relationships. Participants may have up to 3 additional sessions to make up any missed group sessions.

This project is an important and timely pilot study. Previous reviews of interventions suggest there is a gap in effective interventions to treat IPV for those with trauma backgrounds (Cheng et al., 2021; Travers et al. 2021). PARTS1, PARTS2 and PARTS SUD have all demonstrated effective reductions in PTSD symptoms and enhanced emotion regulation and self-related processing (Comeau et al. 2024; Ally et al., submitted; Schuman-Olivier et al., in progress). The protocol's methodology follows previous intimate partner violence studies, incorporating verbal consent and partner inclusion, while employing rigorously implemented informed consent procedures and gold-standard measures to enhance the likelihood of success and publication. By incorporating the Difficulties in Emotion Regulation (DERS) and a WHO-5 for quality of life, we aim to address gaps in understanding the comprehensive factors contributing to intimate partner violence.

Primary Aim

The primary aim of this protocol is feasibility of a live-online version of the PARTS program. Feasibility is defined in two ways: intervention-based feasibility: 70% of participants completing at least 67% (e.g., 8/12) of the first 12 groups, study-protocol feasibility as 67% or more of participants completing week-20 study assessments (H1.1).

Secondary Aims The secondary aims are to examine the overall acceptability of the intervention as measured by the Client Satisfaction Questionnaire (CSQ-8) (Larsen et al., 1979) with a mean score of at least 20 out of a total of 32 (H2.1), and intervention satisfaction as measured by a satisfaction question (would you recommend a friend) obtaining at least a mean of 7 out of 10 (H2.2).

A third secondary aim of the study is to investigate the potential effects of the intervention on the Revised Conflict Tactics Scale (CTS2) (Straus et al., 1996; Chapman & Gillespie, 2019). We hypothesize a risk reduction in physical and psychological violence, with an a priori expectation of obtaining a small to moderate effect size (Cohen's d: 0.2-0.5) from self-reports (H2.3). This effect size aligns with a comparably powered study, Strength at Home, among court-mandated civilians (N=23), which reported moderate effect sizes on CTS2.

ELIGIBILITY:
Inclusion Criteria:

Must be male-identifying or prefer to be in a male-identifying group; Must be a resident of Washington state; Must be court-referred to a treatment program for using violence with an intimate partner; Have sufficient English fluency and literacy skills to understand the consent process, procedures and questionnaires and have the ability to provide written informed consent; Have access to the internet and an electronic device with adequate data capacity; to complete questionnaires online and attend online video conference groups; Must be available and willing to attend 17 out of 20 scheduled online group sessions; and Must be available and willing to complete the online computerized assessments and phone interviews.

Exclusion Criteria:

Insufficiently stable housing or internet connection to be able to join at least 17 sessions; Current participation in another experimental research study; Expected medical hospitalization in the next six months from study enrollment period; Current or expected physical incarceration in the next six months from study enrollment period; Inpatient hospitalization for mental health, substance use, suicide attempt or self-harm within past three months; Inability to participate safely in the study intervention and without disrupting the group (in the opinion of principal investigator OR meeting any of the following criteria) Past year history of a psychotic disorder or clinician confirmed active psychosis assessed by the Structured Clinical Interview for DSM-5 (SCID-5); Bipolar I disorder history or current severe level of mania assessed by the Structured Clinical Interview for DSM-5 (SCID-5); Acute suicidality with intent will be excluded from the study (Structured Clinical Interview for DSM-5 [SCID-5]); High levels of Psychopathy as defined by self-report psychopathy checklist (SRP-4); Self-injurious behavior in past three months will require clinical assessment prior to participation in the program; Acute homicidality with plan and/or intent; Severe personality disorder with clinical history that would suggest potential disruptions within the group as assessed by the Structured Clinical Interview for DSM-5 (SCID-5); and/or Inability to join a group without intoxication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male-identifying participants are eligible to participate.
Enrollment: 24 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | At 12 and 20 weeks
  Intervention-based feasibility: 67% (e.g., 8/12) of participants completing at least 67% (e.g., 8/12) of the first 12 groups, study protocol feasibility as 67% (e.g., 8/12) or more of participants completing week-20 study assessments.

SECONDARY OUTCOMES:
Acceptability of Intervention | At 12 and 20 weeks
  Mean score of 20 on the Client Satisfaction Questionnaire (CSQ-8) general acceptability item.
Intervention Satisfaction | At 12 and 20 weeks
  Mean >7.0 of 10 on willingness to refer a friend on Satisfaction Questionnaire
Revised Conflict Tactics Scale (CTS2) | Change from Baseline to 12 and 20 weeks
  A 78-item self-report scale measuring conflict tactics that are used in relationships

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance Center for Mindfulness and Compassion
Locations (2):
- United States (2):
  - Cambridge Health Alliance Center for Mindfulness and Compassion, Malden, Massachusetts
  - Waterland Counseling, Tumwater, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taft CT, Franz MR, Cole HE, D'Avanzato C, Rothman EF. Examining strength at home for preventing intimate partner violence in civilians. J Fam Psychol. 2021 Sep;35(6):857-862. doi: 10.1037/fam0000732. Epub 2021 Mar 18. PMID 33734765
- [Background] Comeau A, Smith LJ, Smith L, Soumerai Rea H, Ward MC, Creedon TB, Sweezy M, Rosenberg LG, Schuman-Olivier Z. Online group-based internal family systems treatment for posttraumatic stress disorder: Feasibility and acceptability of the program for alleviating and resolving trauma and stress. Psychol Trauma. 2024 Dec;16(Suppl 3):S636-S640. doi: 10.1037/tra0001688. Epub 2024 Jun 27. PMID 38934934